CLINICAL TRIAL: NCT04750421
Title: Transillumination: A Non Invasive Method to Reduce Complications Associated With Facial Injections in Aesthetic Medicine.
Brief Title: Transillumination to Reduce Post-injection Complications in Aesthetic Medicine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helynck, Patrick, M.D. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017-A03325-48
Record Dates: First submitted 2021-02-08; First posted 2021-02-11 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: E05.642.500
Keywords: transillumination; Aesthetic injection; asthetic post-injection complications; hyaluronic acid; Facial injection

STUDY DESIGN:
Intervention Model Description: The random assignment of the right or left side of the face on which the trasnillumination will be used will be done by numbered and sealed envelope.
  Envelopes will be prepared before the start of inclusion. Each envelope will contain a sheet of paper whose contents cannot be guessed when the envelope is closed. Each sheet will be marked either "Left+TL" or "Right+TL". Each envelope will contain a unique code number that will be randomly assigned to each patient after inclusion.
Who Masked: Outcomes Assessor
Masking Description: The operator will guarantee the confidentiality of the part of facial where the trasillumination was used, the assessors will not be aware of the part of the face where the transillumination was used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transillumination Venolux® (Experimental): Transillumination using Venolux was used to visualize veins in the hemiface before hyaluronic acid injections
  Interventions: Device: Transillumination Venolux®
- Comparator group (No Intervention): No vascular exploration methods were used on the other hemiface

INTERVENTIONS:
Device: Transillumination Venolux® — Transillumination Venolux® method was used on the other half of the face before injections to visualize veins.
  Arms: Transillumination Venolux®

SUMMARY:
Transillumination (TL) is a noninvasive technique that appears to allow preliminary detection of superficial vascular structures of the face to avoid intravascular HA injection. The purpose of our study was to test the efficacy of TL in terms of its sensitivity to locate vessels in the areas undergoing treatment and to reduce post-injection vascular complications.

DETAILED DESCRIPTION:
Transillumination was used during the injection of hyaluronic acid to reduce the risk of intravascular injection. For the purpose of randomization, patients were asked to choose a sealed envelope. Inside the envelope was a piece of paper indicating on which side of the face (right or left) the transillumination would be used.

For each filler injection, transillumination was used on one side; on the other side of the face, the injection was administered without the use of any vascular exploration method. After the vessels had been located on the side chosen for the transillumination technique, a skin-marker pencil was used to draw the vascular mapping of the upper part of the face, which in our opinion represented the area most at risk of complications, the middle and the lower parts of the face.

Then ice was applied on both sides of the face for 15 s before to proceed with the injections in order to cause vasoconstriction and to further decrease the risk of an intravascular injection.Transillumination sensitivity for locating the vessels of the face was assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for facial injections of hyaluronic acid

Exclusion Criteria:

* Patients with a history of allergy to a component of hyaluronic acid
* Patients with arteritis (Horton)
* Patients who have had previous facial surgery
* pregnant or nursing patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Number of vessels detected by using transillumination | Before facial injections
  counting the number of vessels detected by using transillumination in relation to the number of existing vessels.

SECONDARY OUTCOMES:
Number of bruises and hematoma | At day 3 after facial injections
  Number of bruises and heamatoma post-injection in in the hemiface where Transillumination is used versus control hemiface

CONTACTS AND LOCATIONS:
Overall Officials: Jean Meningaud, MD.PhD, Principal Investigator — Department of plastic and reconstructive surgery-Henri Mondor Hospital
Locations (1):
- MEZI, Créteil, France